CLINICAL TRIAL: NCT03682003
Title: Hepcidin: a Prognostic Marker of Morbidity and Mortality in Severe Sepsis?
Acronym: HEP-SEPSIS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC13_9906_HEP-SEPSIS
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Severe Sepsis or Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood tests are performed to determine hepcidin, IL-6, CRP, PCT, serum iron, ferritin, transferrin and transferrin saturation
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: blood diagnostic tests — blood tests are performed to determine hepcidin, IL-6, CRP, PCT, serum iron, ferritin, transferrin and transferrin saturation

SUMMARY:
Many biomarkers have been evaluated in sepsis, especially for prognostic purposes, but none has yet been shown to have sufficient sensitivity or specificity for routine use in clinical practice. However, highlighting a biomarker facilitating the evaluation of the severity of sepsis remains relevant in a pathology where survival is largely conditioned by the initiation of an early and adapted treatment. Recent evidence suggests that hepcidin, which is the key hormone for systemic regulation of iron metabolism, may be an interesting prognostic biomarker. The synthesis of this peptide is regulated by the iron stocks of the body, erythropoiesis, but also inflammation. The mechanisms inducing the expression of hepcidin during inflammation are multiple: interleukin-6 (IL-6) in particular, pro-inflammatory cytokine is a strong inducer of hepcidin. In addition, its expression is increased by the effect of lipopolysaccharide via Toll-like receptors . In septic patients, elevated levels of hepcidin or pro-hepcidin have been reported . A new role for hepcidin in the control of inflammatory and / or immune response has recently been reported. Thus, in a model of murine septic shock, the deleterious character of a lack of expression of hepcidin could be demonstrated . In humans, hepcidinemia has been shown to be a predictive factor in the development of immunotolerance in hepatic transplant patients. Hepcidin therefore plays a major role in the regulation of the inflammatory and / or immune response and in particular during sepsis. The investigators therefore hypothesize that hepcidin could be the marker of an adverse prognosis in septic patients expressing this

DETAILED DESCRIPTION:
Many biomarkers have been evaluated in sepsis, especially for prognostic purposes, but none has yet been shown to have sufficient sensitivity or specificity for routine use in clinical practice. However, highlighting a biomarker facilitating the evaluation of the severity of sepsis remains relevant in a pathology where survival is largely conditioned by the initiation of an early and adapted treatment. Recent evidence suggests that hepcidin, which is the key hormone for systemic regulation of iron metabolism, may be an interesting prognostic biomarker. The synthesis of this peptide is regulated by the iron stocks of the body, erythropoiesis, but also inflammation. The mechanisms inducing the expression of hepcidin during inflammation are multiple: interleukin-6 (IL-6) in particular, pro-inflammatory cytokine is a strong inducer of hepcidin. In addition, its expression is increased by the effect of lipopolysaccharide via Toll-like receptors . In septic patients, elevated levels of hepcidin or pro-hepcidin have been reported . A new role for hepcidin in the control of inflammatory and / or immune response has recently been reported. Thus, in a model of murine septic shock, the deleterious character of a lack of expression of hepcidin could be demonstrated . In humans, hepcidinemia has been shown to be a predictive factor in the development of immunotolerance in hepatic transplant patients. Hepcidin therefore plays a major role in the regulation of the inflammatory and / or immune response and in particular during sepsis. The investigators therefore hypothesize that hepcidin could be the marker of an adverse prognosis in septic patients expressing this.

Primary endpoint is to evaluate the prognostic value of plasma hepcidin assayed on admission to intensive care on mortality at D28 in severe sepsis.

Sensitivity of plasma hepcidin assayed at admission to intensive care on mortality at D28 in patients with severe sepsis.

In a first step, a search for the hepcidin threshold value with the best sensitivity and specificity to predict death on D28 will be performed using a receiver operating characteristics (ROC) curve. This threshold value will be used to evaluate the primary endpoint and also determine specificity and positive and negative predictive values.

ELIGIBILITY:
Inclusion Criteria:

* man or woman,
* older than or equal to 18 years, in severe sepsis or septic shock according to the criteria of the American College of Chest Physicians / Society of Critical Care Medicine (ACCP / SCCM),
* no opposition from the patient, a relative or the legal representative

Exclusion Criteria:

* pregnant or lactating woman,
* patient with hemochromatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Man or woman, older than or equal to 18 years, with severe sepsis or septic shock according to the criteria of the American College of Chest Physicians / Society of Critical Care Medicine (ACCP / SCCM),
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of plasma hepcidin assayed at admission to intensive care on mortality at D28 in patients with severe sepsis. | day 28
  Sensitivity of plasma hepcidin assayed at admission to intensive care on mortality at D28 in patients with severe sepsis.

SECONDARY OUTCOMES:
mortality at day 90 | day 90
  mortality at day 90
occurrence of care-related infections as defined by the Center for Disease Control and Prevention during hospitalization | day 90
  occurrence of care-related infections as defined by the Center for Disease Control and Prevention during hospitalization
occurrence of new organ failure (SOFA) or the aggravation of an existing organ failure on seventh day of sepsis | day 90
  occurrence of new organ failure (SOFA) or the aggravation of an existing organ failure on seventh day of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Nesseler, MD, Principal Investigator — Rennes University Hospital